CLINICAL TRIAL: NCT01869959
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY2405319 With 28 Days of Subcutaneous Injections in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2405319 in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 12708; I1K-MC-GLUG (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Results first posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — LY2405319

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo-matching LY2405319 injected subcutaneously (SC) once daily for 28 days.
  Interventions: Drug: Placebo
- 3 mg LY2405319 (Experimental): Participants received 3 milligrams (mg) LY2405319 injected SC once daily for 28 days.
  Interventions: Drug: LY2405319
- 10 mg LY2405319 (Experimental): Participants received 10 mg LY2405319 injected SC once daily for 28 days.
  Interventions: Drug: LY2405319
- 20 mg LY2405319 (Experimental): Participants received 20 mg LY2405319 injected SC once daily for 28 days.
  Interventions: Drug: LY2405319

INTERVENTIONS:
Drug: LY2405319 — Administered SC
  Arms: 10 mg LY2405319; 20 mg LY2405319; 3 mg LY2405319
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study was to evaluate the safety and tolerability of LY2405319. It was given as a daily injection under the skin to participants with type 2 diabetes mellitus (T2DM) for 28 days. This study determined how long the drug stays in the body and how it affects blood sugar levels. After screening, the study lasted about 2 months for each participant. Participants continued their prestudy regimen of diet and exercise alone or in combination with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of T2DM.
* Are on diet and exercise or diet, exercise, and metformin (stable dose of at least 1000 mg/day for at least 60 days) regimen.
* Have a glycosylated hemoglobin A1c (HbA1c) value of 7.0% to 10.0%, inclusive, or are on metformin and an additional oral antidiabetic medication (OAM) with an HbA1c value of 6.5% to 9.5%, inclusive.
* Participants on another OAM in addition to metformin therapy may be randomized if removed from treatment of the other OAM ≥14 days prior to study drug administration and fasting blood glucose is ≥145 mg per deciliter (mg/dL) and ≤270 mg/dL.
* Are females not of child-bearing potential due to surgical sterilization or are postmenopausal.
* Have a body mass index (BMI) ≥25 and ≤40.
* Have clinical laboratory test results within normal reference range for the population.

Exclusion Criteria:

* Use insulin, thiazolidinediones (TZDs), dipeptidyl peptidase (DPP) IV inhibitors, or exenatide during the 3 months prior to screening.
* Have had more than 1 episode of severe hypoglycemia requiring assistance of another person to administer a resuscitative action within 6 months prior to entry into the study or are currently diagnosed with having hypoglycemia unawareness.
* Have had 2 or more emergency room visits or hospitalizations due to poor glucose control in the past 6 months.
* Have any abnormality of the electrocardiogram (ECG) that will, in the opinion of the investigator, impair the ability to measure the QT (a corrected QC [QTc] [Bazett's correction] interval >450 milliseconds [msec] for men and >470 msec for women or a PR interval >220 msec are specifically excluded) or have conduction abnormalities that may confound the QTc analysis.
* Have a personal or family history of long QT syndrome, family history of sudden death, personal history of unexplained syncope within the last year; or use prescription or over-the-counter medications known to prolong the QT or QTc interval.
* Have diastolic blood pressure (DBP) ≥95 millimeters of mercury (mm Hg) and/or systolic blood pressure (SBP) ≥160 mm Hg.
* Have an active or untreated malignancy or have been in remission from a clinically significant malignancy for <5 years.
* Have a history of a transplanted organ.
* Evidence of a significant active, uncontrolled endocrine or autoimmune abnormality, as judged by the investigator, at screening.
* Have a history of human immunodeficiency virus (HIV).
* Have a known allergy to yeast or yeast proteins, history of anaphylaxis with bronchospasm, or atopic dermatitis with chronic urticaria.
* Have any other condition (including known drug or alcohol abuse or psychiatric disorder within the last 6 months) that may preclude the participant from following and completing the protocol.
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (including pancreatitis), hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Are women who are breastfeeding.
* Have had a significant change in weight, defined as a gain or loss of at least 4 kilograms (kg) (9 pounds) in the 90 days prior to randomization.
* Have taken in the 30 days prior to randomization, a medication, herbal product, or nutritional supplement that affects adipose mass or distribution or energy balance.
* Are receiving chronic (>2 weeks) systemic glucocorticoid therapy (excluding topical or inhaled preparations) or have received such therapy within 4 weeks immediately prior to second screening appointment.
* Have current or recent (within the past 3 months) use of gemfibrozil or fenofibrate, niacin, ezetimibe, or bile acid binding resins (for example, cholestyramines). Stable statin therapy of ≥3 months will be allowed.
* Are currently taking central nervous system (CNS) stimulant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cypress, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tustin, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miramar, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 3 mg LY2405319: 3 milligrams (mg) LY2405319 injected SC once daily for 28 days.
- 10 mg LY2405319: 10 mg LY2405319 injected SC once daily for 28 days.
- 20 mg LY2405319: 20 mg LY2405319 injected SC once daily for 28 days.
- Placebo: Placebo-matching LY2405319 injected subcutaneously (SC) once daily for 28 days.
- All Randomized Participants: All participants randomized in the study.
Period: Randomization Period
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo | All Randomized Participants
Started | 0 | 0 | 0 | 0 | 47
Completed | 0 | 0 | 0 | 0 | 46 (One participant discontinued after randomization but did not receive study drug.)
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Period: Treatment Period
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo | All Randomized Participants
Started | 11 | 10 | 15 | 10 | 0 (Participants were randomized to treatment groups for the Treatment Period.)
Received at Least 1 Dose of Study Drug | 11 | 10 | 15 | 10 | 0
Completed | 10 | 8 | 12 | 8 | 0
Not Completed | 1 | 2 | 3 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 3 | 1 | 0
Not completed — Sponsor decision | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- 3 mg LY2405319: 3 mg LY2405319 injected SC once daily for 28 days.
- Total: Total of all reporting groups
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 15 | 10 | 46
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.5 (7.3) | 59.6 (9.2) | 56.9 (10.2) | 58.6 (6.3) | 57.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7 | 6 | 20
  Male | 7 | 7 | 8 | 4 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 10 | 15 | 10 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 11 | 10 | 13 | 10 | 44
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 15 | 10 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: The number of participants with 1 or more SAEs considered by the investigator to be related to study drug administration is reported. SAEs were classified using the Medical Dictionary for Regulatory Activities (MedDRA) 11.0. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through Day 56
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: number of participants
Groups:
- 3 mg LY2405319: Participants received 3 mg LY2405319 injected SC once daily for 28 days.
- Placebo: Participants received placebo-matching LY2405319 injected SC once daily for 28 days.
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 11 | 10 | 15 | 10
number of participants | 0 | 0 | 1 | 0

2. Secondary Outcome: Change From Baseline to Day 28 in Fasting Glucose
Description: Change from baseline to Day 28 in fasting blood glucose is presented. The predose fasting blood glucose measurement on Day 1 served as the baseline value. LS means were calculated using a linear mixed effects model with treatment, day, and treatment times day as fixed effects; baseline as covariate; and participant as a random effect.
Time Frame: Baseline, Day 28
Population: Participants who received at least 1 dose of study drug with evaluable blood glucose data.
Measure: Least Squares Mean (90% Confidence Interval); unit: milligrams per deciliter (mg/dL)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 13 | 8
milligrams per deciliter (mg/dL) | -3.5 [-19.2 to 12.2] | -6.7 [-24.4 to 11.0] | -10.5 [-24.3 to 3.4] | 3.2 [-14.1 to 20.4]

3. Secondary Outcome: 7 Point Self-monitored Blood Glucose (SMBG)
Description: The daily mean of the 7-point SMBG values is presented. Seven-point glucose profiles were measured by participants at baseline and at Week 4. The 7-point SMBG mean on Days -5, -4, or -3 served as the baseline value; the 7-point SMBG mean on Days 24, 25, or 26 served as the Week 4 value. Blood glucose was measured before and 2 hours after each meal and at bedtime.
Time Frame: Baseline (Day -5, -4, or -3) and Week 4 (Days 24, 25, or 26)
Population: All participants who received at least 1 dose of study drug with evaluable 7-Point SMBG data.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 11 | 10 | 15 | 10
mg/dL
  Baseline (Days -6, -5, or -4) | 178.01 (5.95) | 171.13 (5.02) | 183.97 (4.19) | 172.46 (5.33)
  Week 4 (Days 24, 25, or 26) | 171.03 (6.10) | 167.95 (8.09) | 188.52 (7.14) | 177.41 (7.24)

4. Secondary Outcome: Change From Baseline to Week 4 in Glucose Area Under the Curve (AUC)
Description: Change from baseline to Week 4 in glucose AUC during an oral glucose tolerance test (OGTT) is presented. Blood samples were obtained prior to the glucose bolus to 2 hours after administration of the glucose bolus. The AUC measurement on Day -1 served as the baseline value. LS means were calculated using an analysis of covariance model with treatment as fixed effect and baseline as covariate.
Time Frame: Predose and 2 hours postdose (Baseline, Week 4)
Population: All participants who received at least 1 dose of study drug with evaluable glucose AUC data.
Measure: Least Squares Mean (90% Confidence Interval); unit: milligrams*hr per deciliter (mg*hr/dL)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 11 | 8
milligrams*hr per deciliter (mg*hr/dL) | 12.89 [-36.21 to 61.98] | -8.46 [-66.69 to 49.76] | -3.22 [-51.94 to 45.49] | -28.13 [-83.13 to 26.87]

5. Secondary Outcome: Change From Baseline to Week 4 in Insulin Area Under the Curve (AUC)
Description: Change from baseline to Week 4 in insulin AUC during an OGTT is presented. Blood samples were obtained prior to the glucose bolus to 2 hours after administration of the glucose bolus. The AUC measurement on Day -1 served as the baseline value. LS means were calculated using an analysis of covariance model with treatment as fixed effect and baseline as covariate.
Time Frame: Predose and 2 hours postdose (Baseline, Week 4)
Population: All participants who received at least 1 dose of study drug with evaluable insulin (AUC) data.
Measure: Least Squares Mean (90% Confidence Interval); unit: micro International units*hour/mL
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 7 | 12 | 8
micro International units*hour/mL | -10.07 [-20.40 to 0.26] | -10.37 [-23.11 to 2.36] | -15.66 [-25.11 to -6.21] | -17.98 [-29.54 to -6.42]

6. Secondary Outcome: Change From Baseline to Week 4 in C-peptide Area Under the Curve (AUC)
Description: Change from baseline to Week 4 in C-peptide AUC during an OGTT is presented. Blood samples were obtained prior to the glucose bolus to 2 hours after administration of the glucose bolus. The AUC measurement on Day -1 served as the baseline value. LS means were calculated using an analysis of covariance model with treatment as a fixed effect and baseline as covariate.
Time Frame: Predose and 2 hours postdose (Baseline, Week 4)
Population: All participants who received at least 1 dose of study drug with evaluable C-peptide AUC data.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms*hours/milliliter (ng*hr/mL)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 12 | 8
nanograms*hours/milliliter (ng*hr/mL) | -0.61 [-1.58 to 0.36] | 0.07 [-1.03 to 1.17] | -1.39 [-2.27 to -0.51] | -1.59 [-2.66 to -0.51]

7. Secondary Outcome: Change From Baseline to Day 28 in Fasting Lipid Profile
Description: Change from baseline to Day 28 in fasting lipids, including cholesterol, low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), and triglycerides is presented. The predose measurement for each variable on Day 1 served as the baseline value. LS means were calculated using a linear mixed effects model with treatment, day, and treatment times day as fixed effects; baseline as covariate; and participant as a random effect.
Time Frame: Baseline, Day 28
Population: All participants who received at least 1 dose of study drug with evaluable fasting lipid (ie, cholesterol, LDL-C, HDL-C, and triglyceride) data.
Measure: Least Squares Mean (90% Confidence Interval); unit: milligrams per deciliter (mg/dL)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 13 | 8
milligrams per deciliter (mg/dL)
  Cholesterol (n=10, n=8, n=13, n=8) | 3.9 [-6.8 to 14.6] | -32.5 [-44.5 to -20.6] | -31.4 [-40.7 to -22.0] | -1.3 [-13.0 to 10.4]
  LDL-C (n=10, n=8, n=13, n=7) | -0.1 [-10.5 to 10.3] | -26.8 [-38.6 to -14.9] | -24.2 [-33.3 to -15.1] | -0.8 [-13.1 to 11.5]
  HDL-C (n=10, n=8, n=13, n=8) | 10.6 [7.1 to 14.0] | 10.2 [6.3 to 14.1] | 9.1 [6.0 to 12.1] | -0.8 [-4.7 to 3.1]
  Triglycerides (n=10, n=8, n=13, n=8) | -38.5 [-62.9 to -14.1] | -81.0 [-107.3 to -54.8] | -84.4 [-105.0 to -63.8] | 6.8 [-21.2 to 34.9]

8. Secondary Outcome: Change From Baseline to Day 28 in Body Weight
Description: Change from baseline to Day 28 in body weight is presented. The predose body weight measurement on Day 1 served as the baseline value. LS means were calculated using a linear mixed effects model with treatment, day, time, and treatment times time, treatment times day, and treatment times day times time were fixed effects; baseline as covariate; and participant as a random effect.
Time Frame: Baseline, Day 28
Population: All participants who received at least 1 dose of study drug with evaluable body weight data.
Measure: Least Squares Mean (90% Confidence Interval); unit: kilograms (kg)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 13 | 8
kilograms (kg) | -0.7 [-1.6 to 0.3] | -1.8 [-2.9 to -0.6] | -1.5 [-2.3 to -0.7] | -0.2 [-1.3 to 0.8]

9. Secondary Outcome: Change From Baseline to Day 28 in Adiponectin
Description: Change from baseline to Day 28 in adiponectin is presented. The predose adiponectin measurement on Day 1 served as the baseline value. LS means were calculated using a linear mixed effects model with treatment, day, treatment times day as fixed effects, baseline as covariate, and participant as random effect.
Time Frame: Baseline, Day 28
Population: All participants who received at least 1 dose of study drug with evaluable adiponectin data.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 12 | 8
nanograms per milliliter (ng/mL) | 1850.7 [405.1 to 3296.3] | 2907.1 [1289.1 to 4525.1] | 5648.6 [4345.2 to 6952.1] | 458.3 [-1165.1 to 2081.6]

10. Secondary Outcome: Change From Baseline to Day 28 in C-Reactive Protein
Description: Change from baseline to Day 28 in C-reactive protein is presented. The predose C-reactive protein measurement on Day 1 served as the baseline value. LS means were calculated using a linear mixed effects model with treatment, day, and treatment times day as fixed effects; baseline as covariate; and participant as random effect.
Time Frame: Baseline, Day 28
Population: All participants who received at least 1 dose of study drug with evaluable C-reactive protein data.
Measure: Least Squares Mean (90% Confidence Interval); unit: milligrams per liter (mg/L)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 13 | 8
milligrams per liter (mg/L) | -0.6 [-2.5 to 1.3] | 0.3 [-1.8 to 2.4] | 0.0 [-1.6 to 1.7] | 0.4 [-1.8 to 2.5]

11. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Time Curve (AUC) of LY2405319
Description: AUC for LY2405319 is presented. Data represent AUC for 1 dosing interval at steady state. Blood samples were collected predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, and 48 hours postdose on Day 28.
Time Frame: Predose through Day 28 (48 hours postdose)
Population: All participants who received at least 1 dose of study drug with evaluable AUC of LY2405319 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319
Number analyzed (Participants) | 11 | 10 | 15
nanograms*hours/milliliter (ng*hr/mL) | 409 (26.0) | 1520 (38.9) | 3410 (35.1)

12. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY2405319
Description: Cmax of LY2405319 is presented. Blood samples were collected predose and at 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 24, and 48 hours postdose on Day 28.
Time Frame: Predose through Day 28 (48 hours postdose)
Population: All participants who received at least 1 dose of study drug with evaluable Cmax of LY2405319 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319
Number analyzed (Participants) | 10 | 8 | 12
nanograms per milliliter (ng/mL) | 39.9 (34.7) | 105 (62.9) | 247 (58.8)

13. Secondary Outcome: The Number of Participants With Anti-LY2405319 Antibodies
Description: The number of participants that tested positive for anti-LY2405319 antibodies is presented.
Time Frame: Day 1 through Day 56
Population: All participants who received at least 1 dose of study drug with evaluable anti-LY2405319 antibody data.
Measure: Number; unit: number of participants
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 11 | 10 | 15 | 10
number of participants | 6 | 8 | 13 | 2

14. Secondary Outcome: Change From Baseline to Day 28 in Eating Inventory for Cognitive Restraint of Eating, Disinhibition, and Hunger
Description: Change from baseline to Day 28 in Eating Inventory (EI) subscales are presented. The EI is a 51-item inventory that measures dietary restraint (the cognitive intention to restrict energy intake; scores range from 0 to 21), disinhibition (the tendency to episodically overeat, often in response to external cues; scores range from 0 to 16), and perceived hunger (scores range from 0 to 14). A low score indicates a low exhibition of behavior and a high score indicates a high exhibition of behavior. The measurement for each variable obtained on Day -2 served as the baseline value. LS means were calculated using an analysis of covariance model with treatment, day, and treatment times day as fixed effects, and baseline as covariate.
Time Frame: Baseline, Day 28
Population: All participants who received at least 1 dose of study drug with evaluable EI data.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 12 | 8
units on a scale
  Cognitive restraint of eating | -1.10 [-2.68 to 0.48] | -0.35 [-2.09 to 1.39] | -0.27 [-1.71 to 1.17] | -2.99 [-4.73 to -1.25]
  Disinhibition | 0.34 [-0.67 to 1.34] | 0.04 [-1.06 to 1.15] | -1.59 [-2.47 to -0.70] | 0.04 [-1.06 to 1.14]
  Hunger | 1.00 [-0.32 to 2.32] | 2.05 [0.59 to 3.50] | 0.53 [-0.65 to 1.70] | 0.29 [-1.16 to 1.73]

15. Secondary Outcome: Change From Baseline to Day 28 in the Food Preference Questionnaire (FPQ) Score
Description: The table below represents the change from baseline in FPQ total score. The FPQ was administered to assess overall preference for foods of different macronutrient contents utilizing a macronutrient self-selection paradigm. Participants rated their preference on a range from 1 to 9 with 1 (dislike extremely) to 9 (like extremely) for a battery of 72 commonly consumed foods with fat content varying significantly in sugar, complex carbohydrates, and protein. The total score was calculated by averaging preference scores of 72 items. A low mean score of 1 to 9 scale indicate a low preference for the foods listed and a high mean score indicate a high preference for the foods listed. The FPQ measurement on Day -2 served as the baseline value. LS means were calculated using an analysis of covariance model with treatment, day, and treatment times day as fixed effects, and baseline as covariate.
Time Frame: Baseline, Day 28
Population: All participants who received at least 1 dose of study drug with evaluable FPQ data.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 12 | 8
units on a scale | -0.06 [-0.73 to 0.61] | -0.43 [-1.15 to 0.29] | -0.77 [-1.30 to -0.24] | 0.74 [0.09 to 1.40]

16. Secondary Outcome: Change From Baseline to Day 28 in The Patient Health Questionnaire (PHQ-9) Score
Description: Change from baseline to Day 28 in the PHQ-9 total score is presented. Participants were asked to score the severity of depressive symptoms over the last 2 weeks. Items were scored 0 (not at all), 1 (several days), 2 (half of the days), or 3 (nearly every day). The total PHQ-9 score is the sum of the score for each item and range from 0 to 27. A score of 0 means low depression severity and a score of 27 means high depression severity. Depression severity will be given a quality rating based on the total PHQ-9 score, as follows: None (0-4); Mild (5-9); Moderate (10-14); Moderately severe (15-19); and Severe (20-27). The PHQ-9 measurement obtained on Day -2 served as the baseline value. LS means were calculated using an analysis of covariance model with treatment, day, and treatment times day as fixed effects, and baseline as covariate.
Time Frame: Baseline, Day 28
Population: All participants who received at least 1 dose of study drug with evaluable PHQ-9 data.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Number analyzed (Participants) | 10 | 8 | 12 | 8
units on a scale | 1.26 [-0.71 to 3.24] | -0.50 [-2.83 to 1.82] | 1.82 [0.08 to 3.56] | 2.57 [0.43 to 4.71]

ADVERSE EVENTS:
Arm/Group | 3 mg LY2405319 | 10 mg LY2405319 | 20 mg LY2405319 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10 | 2/15 | 1/10
Other Adverse Events (participants affected / at risk) | 7/11 | 8/10 | 11/15 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg LY2405319 (N=11) | 10 mg LY2405319 (N=10) | 20 mg LY2405319 (N=15) | Placebo (N=10)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3 mg LY2405319 (N=11) | 10 mg LY2405319 (N=10) | 20 mg LY2405319 (N=15) | Placebo (N=10)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Application site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (3) | 6 (39) | 7 (46) | 2 (2)
Injection site haemorrhage (General disorders) | 0 (0) | 5 (7) | 6 (11) | 3 (6)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Injection site inflammation (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Injection site irritation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 3 (6) | 1 (2) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcium increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (2)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (7) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days